CLINICAL TRIAL: NCT00919087
Title: Evaluating Ventricular Events With Adherent Patient Monitoring Study
Brief Title: Non Invasive Arrhythmia Detection in Hospital Settings
Acronym: EVE
Status: Completed | Type: Observational
Sponsor: Corventis, Inc. (Industry)
Responsible Party: Madhuri Bhat, VP Regulatory and Clinical affairs, Corventis
Other Study IDs: COR-2009-002
Record Dates: First submitted 2009-06-10; First posted 2009-06-12 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2010-02

CONDITIONS: Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Avivo System — Non invasive external monitoring deive
  Other Names: external monitoring systems

SUMMARY:
This is a prospective, single center, non-randomized study to evaluate the arrhythmia detection performance during ventricular events.

DETAILED DESCRIPTION:
The system will continuously monitor the patient's cardiac activity which will be compared to standard telemetry system.

ELIGIBILITY:
Inclusion Criteria:

* Is female or male, 18 years of age or older
* Undergoing ICD implant with ventricular arrhythmia induction OR undergoing EP study with ventricular arrhythmia induction

Exclusion Criteria:

* Is participating in another clinical study that may confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: electrophysiology (EP) study or implantable cardioverter defibrillator (ICD) implant Patients
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imad Libbus, PhD, Study Director — Corventis, Inc.